CLINICAL TRIAL: NCT02464423
Title: Improving Adherence Among HIV+ Rwandan Youth: A TI-CBTe Indigenous Leader Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hektoen Institute for Medical Research (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HD074977 (NIH)
Record Dates: First submitted 2015-04-10; First posted 2015-06-08 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Usual care: WE-ACTx For Hope and CHUK offer a host of services for HIV+ young people, and these will represent the "usual care" condition for the study. Both clinics provide adolescent-friendly environments with multidisciplinary teams that offer weekly or monthly support groups, peer education, medical services, mental health screenings, sports activities, HIV and health education sessions, and outreach to parents and guardians. The services youth in the "usual care" condition receive will be carefully tracked.
- Treatment (Active Comparator): Culturally-adapted, trauma-informed cognitive behavioral therapy (TI-CBT) intervention: The components of the TI-CBT include a) psychosocial health education b) relaxation training c) cognitive restructuring d) adherence barriers e) caregiver psycho-education. The TI-CBTe will be administered in groups of 8-10 weekly for 2 hours for 3 Sundays each month over 2 months. Two IYL will co-lead each intervention, and two IYL will rate fidelity.
  Interventions: Behavioral: Trauma-Informed Cognitive Behavioral Therapy enhanced (TI-CBTe)

INTERVENTIONS:
Behavioral: Trauma-Informed Cognitive Behavioral Therapy enhanced (TI-CBTe)
  Arms: Treatment

SUMMARY:
Like most of sub-Saharan Africa, Rwandan youth are the epicenter of the AIDS epidemic, accounting for 40% of new infections. Antiretroviral (ART) adherence is a global health priority, but Rwandan youth are more than twice as likely to be on second line therapy than adults, and with a median population age of 18.7 years old, adherence is essential for Rwanda's future. Resources to provide youth-centered medical and psychosocial care are limited in Rwanda, and young people with HIV face many obstacles to adherence, namely the long-term consequences of genocide, depression, and gender-based violence, as well as logistical issues, negative attitudes, and insufficient parent/caregiver support. Preliminary data underscore the utility of culturally-adapted, trauma-informed cognitive behavioral therapy (TI-CBT) in reducing depression and traumatic distress among youth and adults in Rwanda. This project proposes a 2-arm randomized controlled trial (RCT) to test and compare the efficacy of adherence-enhanced Trauma Informed Cognitive Behavioral Therapy (i.e., TI-CBTe) to usual care in increasing ART adherence among Rwandan youth from two clinics caring for the largest number of youth with HIV in Rwanda. This proposal answers a compelling need for innovative programs to increase ART adherence among HIV+ youth. If effective, the study will build Rwanda's capacity to provide much needed services; and, involvement by the Rwanda Biomedical Center will ensure wide dissemination.

DETAILED DESCRIPTION:
This study proposes a 2-arm, RCT to test and compare adherence-enhanced Trauma Informed Cognitive Behavioral Therapy (TI-CBTe) to usual care on ART adherence among HIV+ Rwandan youth. Based on a well-grounded theoretical framework, TI-CBTe blends a culturally adapted empirically-supported intervention (TI-CBT) with strategies to increase ART adherence by reducing depression, trauma, and gender based violence (GBV). 350 HIV+ 14-21 year olds will be randomly assigned to TI-CBTe or usual care and the intervention will be delivered in small groups of 8 - 10 over eight consecutive Sundays. Adult caregivers (where available) will participate in two sessions to address adherence support for youth. Caregivers and youth will complete assessments at baseline, 6 and 12 months. Consistent with the Indigenous Leader Outreach Model (ILOM), HIV+ young adults who are > 95% ART adherent will be trained to deliver TI-CBTe. An intent-to-treat analysis will be used and a combination of regression techniques and other inferential statistical tests for contrasting means and proportions. Treatment effects on adherence and mediators for youth participants will be examined, as well as indigenous youth leaders. Treatment outcomes will be analyzed using logistic and linear multiple regression models examining effects at 6- and 12- months separately, as well as a combined model with random effects for repeated measurements across time.

Participants will be recruited from two clinics: WE-ACTx For Hope and Central University Hospital of Kigali (CHUK), which are the primary providers of HIV care for infected adolescents, and both have long-standing relationships with the community. Youth and caregivers will be invited to meet with research staff if they are interested to inform them about the project and request permission to be contacted by the research team. The assent/consent forms will be reviewed with IYL, youth and caregivers, and trained staff will administer questionnaires and interviews. Both sites have a staff psychologist who will provide clinical backup in cases of mental health distress. Consent/assent forms will state the exceptions to confidentiality, and where a youth reports child abuse or neglect or suicidal ideation or attempts, the psychologist will be consulted. Indigenous youth leaders (IYL), youth and caregivers will each complete the baseline and two follow-up assessments. A month before follow-ups, IYL, youth and caregivers will be contacted to request their participation in the next wave of data collection. Transportation will be offered and interviews will be conducted at the clinics in a confidential location.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* 14-21 years old
* seeking HIV care and treatment
* enrolled in support groups at CHUK or We-ACTx For Hope
* able to understand the informed consent process.

Exclusion Criteria:

* are unable to understand the consent/assent process
* do not speak Kinyarwanda (all instruments will be translated and back-translated)
* are not HIV+
* received an HIV diagnosis in the past week

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 731 (Actual)
Dates: Start 2013-01; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
ART Adherence Behavior Composite Self Report | Up to 12 months
  ART adherence behavior measured by self report. Report is a composite of several validated internationally used measures (7 day recollection, 6 month judgement of overall adherence and appreciation of stopping medications).

SECONDARY OUTCOMES:
Health Care Utilization (Number of Clinic Visits) | Up to 12 months
  Track number of mental health and support services visits by youth in both treatment arms.

OTHER OUTCOMES:
HIV/AIDS/Sexually Transmitted Infection (STI)-risk | Up to 12 months
  The AIDS-Risk Behavior Assessment (ARBA) measures self-reported sexual behavior and drug use.

CONTACTS AND LOCATIONS:
Overall Officials: Mardge Cohen, MD, Principal Investigator — We-ACTx; Sabin Nsanzimana, MD, Principal Investigator — Rwanda Biomedical Centre; Geri Donenberg, PhD, Principal Investigator — University of Illinois Chicago
Locations (2):
- Rwanda (2):
  - Cental University Hospital of Kigali - CHUK, Kigali
  - WE-ACTx for Hope, Kigali

REFERENCES:
- [Derived] Donenberg GR, Fitts J, Ingabire C, Nsanzimana S, Fabri M, Emerson E, Remera E, Manzi O, Bray B, Cohen MH. Results of the Kigali Imbereheza Project: A 2-Arm Individually Randomized Trial of TI-CBT Enhanced to Address ART Adherence and Mental Health for Rwandan Youth Living With HIV. J Acquir Immune Defic Syndr. 2022 May 1;90(1):69-78. doi: 10.1097/QAI.0000000000002911. PMID 35013089